CLINICAL TRIAL: NCT07129096
Title: Treatment of Temporomandibular Pain and Disorders With Applied Relaxation Trained Using a Web Application- a Randomized Controlled Trial
Brief Title: Digitally Trained Applied Relaxation for Treatment of Temporomandibular Pain
Acronym: RCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: University of Eastern Finland (Other); Tampere University (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Kirsi Sipilä, Professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2025-06-19; First posted 2025-08-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: randomized controlled trial
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Applied relaxation treatment (Experimental): web-based training for applied relaxation
  Interventions: Behavioral: Applied Relaxation
- Occlusal splint (Active Comparator): Occlusal splint treatment (traditional treatment)
  Interventions: Device: Occlusal splint

INTERVENTIONS:
Behavioral: Applied Relaxation — Applied relaxation method developed by psychologists from progressive relaxation is used. The method is trained using a web application (Relappy.app), which contains step-by-step instructions with self-instructed exercises and exercise diaries, in which the examinee records his/her level of tension before and after the exercise (on a scale of 0-100, where 0 means a completely relaxed state, 50 a normal state (neither relaxed nor tense) and 100 maximum tenseness.
  Arms: Applied relaxation treatment
Device: Occlusal splint — The splint group is treated with occlusal splint, which is a conventional treatment method in cases where the implementation of information and self-care methods has not given a sufficient treatment response. The splint is prepared for night use and controlled according to the usual protocol.
  Arms: Occlusal splint

SUMMARY:
Temporomandibular disorders (TMD) are common musculoskeletal pain conditions related to masticatory muscles and temporomandibular joints. Applied relaxation (AR) is a self-management method widely used and tested for treatment of various psychological and somatic conditions, including musculoskeletal pain and other chronic pain conditions. AR is trained step-by-step on a 6-week program under guidance of health care professional. For training of AR, a web application (Relappy) has been developed in University of Oulu, Finland.

The aim of the project is to test the Relappy for training of AR. At first, Relappy is tested by volunteers (n=26). The randomized controlled trial on TMD patients evaluates the effectiveness of web application-based AR training on TMD pain symptoms, psychosocial burden, sleep quality and autonomic nervous system (ANS) activity. The study sample includes TMD patients (n=124) from Finnish Student Health Service in Oulu and Turku units. They are randomly assigned to 2 treatment groups: AR group (trained by AR web application) and stabilization splint group (traditional treatment). TMD pain, body pain, psychosocial symptoms and sleep problems are assessed with validated questionnaires at baseline and at 6-week, 3- month and 1-year follow-up points. The patients also use a digital sleep diary application. Additionally, ANS activity is measured from patients in Oulu before treatment and 3 months weeks and 1 year after baseline. In the analyses, the variables are compared between treatment groups. The present project also includes preparing of the commercialization, aiming to develop the Relappy for wider target groups of pain patients and public use, regardless of time and place of use.

The project has many societal and economic impacts. It can be expected that when actively trained, web application for AR will offer a cost-efficient self-management method to relieve TMD pain, body pain, and other stress-related symptoms and thus improve general well-being. It is expected to reduce healthcare costs and treatment burden and promote sustainability.

DETAILED DESCRIPTION:
Background and significance More than 30% of people worldwide suffer from chronic pain, which causes human suffering for the individual and burdens the society financially. Musculoskeletal diseases are the most functionally impairing diseases in Europe. Masticatory muscle/jaw joint pains and dysfunctions (temporomandibular disorders, TMD) located in the face and head area are the second most common musculoskeletal pain conditions after low back pain. Various biopsychosocial risk factors, such as stress, depressive symptoms, anxiety, and sleep problems are related to chronic pain, including TMD pain. On the other hand, treating sleep disorders can also alleviate pain. Psychological stress and disturbances in the regulation of the pain mechanism related to chronic pain can manifest as dysfunction in the autonomic nervous system (ANS) activity. Compared to healthy people, TMD patients have impaired response of the ANS activity as indicated by higher heart rate, lower heart rate variability and lower baroreflex. Oral prafunctions, such as awake bruxism (tooth clenching during awakefulness) are also common in individuals with TMD and may share common psychosocial background factors with TMD, such as somatic symptoms, depression and anxiety.

Treatment of TMD aims to relieve pain and improve function. Usual treatment methods are counselling and guidance, muscle exercises, manual therapy, and occlusal splint therapy. Motivation and activation of the patient instead of the patient "receiving" passive treatment is important. Structured self-care methods should also be developed and evaluated considering cost-effectiveness. The Current Care Guidelines of pain emphasize the use of patient's own coping strategies. Relaxation training is mentioned as one of these methods, in addition to information, cognitive coping methods, and physical exercises.

Applied relaxation (AR) is a self-management method developed on the basis of Jacobson's progressive relaxation. The method is based on step-by-step training during a six-week programme where the person gradually learns the skill of relaxing his/her body in about 30 seconds. Learning this skill can be compared, for example, to learning to ride a bicycle, where the skill eventually becomes automatic.

AR has been used in treatment of various psychological and somatic conditions, such as anxiety disorders, panic disorders, dental fear, stress problems, gynaecological pain problems, tinnitus, musculoskeletal pains, as well as TMD symptoms, based on a previous randomised controlled trial. As a method that activates the patient and is easy to use independently, AR has several advantages compared to other coping or imagination-based methods. The patient is guided to control his/her reactions and sensations of the ANS by relaxing the body and/or muscle groups. The time needed for relaxation gradually decreases from 20 minutes to less than a minute and transforms from conscious to unconscious through active practice. This method is generally used in the treatment of chronic pain, mostly in specialised medical care units in group meetings under the guidance of a health care professional. There is a need for digital technology for training of AR, which could target it at a wider group of patients.

For training of AR a web application, named Relappy, was developed in University of Oulu and Oulu University Hospital in company collaboration as well as using the expertise on the field of psychology. The Relappy contains instructions, self-instructed exercises and exercise diaries for independent training of AR.

The aim of this randomized controlled study (RCT) is to evaluate the effect of digitalised AR training (by using Relappy) on TMD pain and comorbid symptoms, such as other musculoskeletal pain, psychological symptoms (depression/ anxiety symptoms, unspecific physical symptoms, sleep problems), and oral parafunctions (including sleep and awake bruxism).

Based on the previous knowledge, it can be hypothesized that digitalized AR training relieves TMD pain, other musculoskeletal pain, psychosocial burden, stress-related symptoms as well as oral parafunctions more effectively as compared to "traditional TMD treatment". It can also be seen as lowering of the sympathetic activity in ANS parameters.

As a high-quality clinical study, this RCT trial generates new knowledge for cost-effective treatment of TMD, musculoskeletal pain symptoms, and stress-related symptoms. It emphasizes the patient´s own responsibility and activation, instead of mere "doctor´s tricks", which mostly do not have any far-reaching effects. The study will also offer tools for prevention of stress-related symptoms/ diseases and thus support the welfare and healthcare.

Impact The present high-quality RCT study generates new knowledge on the effectiveness of self-care methods for treatment of TMD and its comorbid symptoms, such as other musculoskeletal pain, psychosocial burden and sleep problems. The merit also comes from that comorbid symptoms are evaluated besides TMD pain, thus considering the larger view of the patient´s condition. It also gives additional value by generating new, clinical-based science, as these is still relatively low number of RCTs in the field of TMD and self-care procedures in pain management.

Training of AR using the Relappy gives many benefits for the users. They get important knowledge about their general health and themselves. This knowledge helps users to achieve positive changes in their lives and to cherish their healthy life habits, which have further effects on working life, relationships and self-confidence. Well-being will improve, and the burden for health care will decrease as the users can themselves do treatment/preventive actions. Although the traditional group meetings of AR have their advantages, digitalisation would offer an efficient and flexible use of the method, also considering the accessibility of the treatment, the patient's time use, healthcare resources and sustainable development (traveling to the office decreases). This would also promote equality, as training of AR can be offered to larger patient groups and non-patients. The online application would enable the AR training to be more widely available, both geographically and temporally, and would reduce the burden on the nursing staff.

Based on the previous randomised controlled trial, AR (trained as traditional group meeting) was more effective in promoting comprehensive wellbeing as compared to occlusal splint treatment. Therefore, it is expected that if actively used, Relappy would achieve corresponding results; not only relieving local TMD pain but also decreasing other body pain and psychosocial burden. Improvement of the quality of sleep is also expected.

The digitally trained AR is expected to give several positive outcomes for individuals suffering from chronic pain by decreasing pain-related disability, improving sleep quality, and promoting psychological well-being. This method can be used in addition to other treatments as part of comprehensive, individualised treatment. The use of Relappy could also prevent the onset of symptoms and development of chronic pain conditions when used regularly and specifically in various stress-related situations. The AR method has no adverse effects.

If shown to be effective, this method can be adopted by clinicians as part of comprehensive, individual treatment of pain patients. The results of the project will be disseminated to the stakeholders, i.e., the wellbeing services counties in Finland.

The expected economic impact is the reduction of healthcare costs by avoiding invasive treatments and medications and by decreasing the number of visits. In Finland, 7-9% of the population need TMD treatment, corresponding to 440,000 people. In the latest comprehensive Healthy Finland Survey in 2023 the preliminary results showed that 7% of Finnish adults (aged 20 years or older) reported of using occlusal splint, corresponding 313,600 people (yet unpublished data). The total cost of one occlusal splint as "traditional" treatment for TMD is approximately 500 euros (including cost for dental technician and salaries for health care personnel), resulting in costs of 156.8 million euros. The occlusal splint may at best be used for a few years and must be renewed thereafter. AR training with the aid of Relappy is expected to replace the occlusal splint at least to some extent, roughly estimating 25% of those in need for treatment, corresponding 96,259 people. When regularly trained, the possible benefit for the patients would be long-lasting.

Besides TMD, Relappy can be used for other pain conditions as well. In 2022, musculoskeletal diseases were the most common reason to seek treatment in health care and also the most common cause of disability retirement. In Finland, musculoskeletal symptoms and diseases cost several billion euros annually. Direct costs include treatment visits, medications, and rehabilitation. Indirect costs are caused by sick leaves, decreased productivity, and unemployment. In 2022 in Finland, musculoskeletal diseases caused costs amounting to 235.2 million euros due to sick leaves and 346.6 million euros due to retirement. The costs of medications due to musculoskeletal diseases were 64.2 million euros. The use of Relappy is expected to decrease these costs, offering safe, non-medication treatment.

Implementation

Preliminary data Before RCT, Relappy was tested by volunteers in a pilot study. The study participants were recruited by e-mail advertisement from the staff and dental students in University of Oulu and Eastern Finland. Feedback on the use of the online service was collected from the participants. In addition, the research subjects answered the same questionnaires as the patients of the clinical study (see section Clinical study). The subjects' self-assessed degree of relaxation before and after the exercises is saved on the server.

Altogether 54.5% responders (n=26) had noted positive changes in their well-being. Based on the questionnaire, the total number of physical symptoms (p=0.017, ANOVA test) and body pain sites (p=0.006) decreased after Relappy training, as compared to the baseline. A tendency of decrease in depression symptoms was also noted (p=0.059). There was also a tendency for improvement of distinct sleep parameters (sleep onset duration, sleep duration), based on the sleep diary Oneiros.

Clinical study The goal of the present study is to evaluate the effectiveness of Relappy on TMD pain symptoms, psychosocial burden factors, sleep quality and oral parafunctions in TMD pain patients of the Finnish Student Health Service (health care units in Oulu and Turku) and two well-being servives counties in Finland (North Ostrobothnia, Oulu, and North Savo, Kuopio), based on a clinical randomised controlled trial (RCT).

The sample is selected from patients who seek treatment due to TMD-related pain symptoms. Subjects are randomly divided into two treatment groups, the AR group and the stabilization splint group. Allocation into groups is performed using a randomization method performed by a computer program.

The exclusion criteria are as follows:

* serious general illnesses such as rheumatism, schizophrenia or other serious mental illness
* pregnancy

The inclusion criteria are as follows:

• presence of TMD pain diagnosis (myalgia, myofascial pain with referral, arthralgia and/or headache attributed to TMD), based on a validated, international Diagnostic Criteria for TMD Axis I criteria

The sample size was calculated using a power calculation. It has been estimated that the difference between two NRS (Numerical Rating Scale, 0-10) points is calculated as a clinically significant pain reduction in the assessment of pain intensity. A mean difference of 2 points (SD 3.5) between groups (at 80% power, statistical significance p<0.05) is obtained with a sample size of 39 patients in each group (78 in total). Added to this is the estimated number of dropouts, which in the previous study was 58 % at 1-year follow-up, resulting in total number of 124 (62 patients/group).

All patients participate in TMD treatment program, where they at first receive information and self-care instructions. If TMD symptoms persist, the patients undergo a new evaluation of the need for treatment. If the patient is willing to participate in the study, he/she will be referred to a clinical examination based on DC/TMD protocol, including symptoms questionnaire and clinical examination (measurement of mandibular range of motion, registration of joint sounds, palpation of masticatory muscles and jaw joints, and registration of mandibular movement pain). Before treatment, the patients fill in a Webropol -based questionnaire inquiring the following information: general diseases, medications, height and weight, use of psychoactive substances (alcohol, tobacco, snuff, drugs), pain symptoms in other parts of the body, psychosocial symptoms and psychological burden are assessed with the validated DC/TMD Axis II questionnaires concerning non-specific physical symptoms (Patient Health Questionnaire-15, PHQ-15), depressive symptoms (PHQ-9), anxiety symptoms (General Anxiety Disorder-7, GAD-7, TMD pain-related intensity/ interference (Graded Chronic Pain Scale, GCPS2.0), oral parafunctions (Oral Behaviors Checklist, OBC). Sleep quality is measured with the validated SCI (Sleep Condition Indicator) questionnaire and with a digital sleep diary during the intervention using a mobile application (Oneiros sleep diary, Oneiros Therapies Oy Ltd). In the follow-up, the sleep diary is filled in for 2 weeks before the treatment and for 2 weeks before the 3-month and 12-month follow-up points.

Treatment of the groups:

1. The splint group is treated with occlusal splint, which is a conventional treatment method in cases where the implementation of information and self-care methods has not given a sufficient treatment response. The splint is prepared for night use and controlled according to the usual protocol.
2. For the second group, the AR method developed by LG Öst from progressive relaxation is used, trained using the Relappy. The web application Relappy contains step-by-step instructions with self-instructed exercises and exercise diaries, in which the examinee records his/her level of tension before and after the exercise (on a scale of 0-100, where 0 means a completely relaxed state, 50 a normal state (neither relaxed nor tense) and 100 maximum tenseness.

In the follow-up questionnaires, both groups fill out the Webropol questionnaires (body pain symptoms, PHQ-15, PHQ-9, GAD-7, GCPS2.0, OBC and SCI) at the 6-week, 3-month and 1-year follow-up points. The Relappy contains links to the questionnaires before starting the relaxation program and after 6 weeks. Otherwise, the links to the questionnaires will be sent by e-mail. In the 6-week follow-up, the relaxation group will also be asked for feedback on the use of the for further development.

Measurements of autonomic nervous system (ANS) activity A sub-sample (n=31) is formed from the subjects from Oulu for whom measurements of ANS activity are made before the treatment and 3 months and 1 year after beginning of the treatment. Heart rate variability, continuous blood pressure and baroreflex sensitivity are measured at the University of Oulu, Biomedical and Internal medicine Research Unit. Body composition is measured (InBody 720, InBody Co. Korea), and after 5 minutes of rest, an ECG (MAC 5500 HD ECG System, GE Healthcare, USA), continuous blood pressure from a finger (Nexfin, BMEYE Medical Systems, the Netherlands) and respiratory rate with a breathing belt (PneumoTrace, AD Instruments, Sydney, Australia) are recorded. The results are analysed for short-term heart rate variability, blood pressure variability and baroreflex sensitivity using software developed at the University of Oulu. After this, the subjects are fitted with EKG (electrocardiogram) Holter equipment and a 24-hour EKG is measured (Faros 360, Bittium, Oulu, Finland). From this, the 24-hour heart rate interval variation over the entire measurement period and separately day (10:00-21:00) and night (01:00-05:00) values are analysed.

Statistical analysis of the data The data is saved to the SSPS Statistics 28.0 program. In the statistical analyses, the following variables are compared between the groups at different time points: pain intensity (NRS), pain intensity/ interference (GCPS2.0), number of pain areas of the body and sum variables of PHQ-9, PHQ-15, GAD-7 and SCI. The digital sleep diary automatically calculates key sleep parameters weekly (sleep efficiency, falling asleep delay, wakefulness during the night, refreshing sleep, sleep duration and number of naps; minimum, average and maximum). These parameters are compared between the groups at the registered time points. In addition, variables of ANS activity are compared between groups at different time points. The comparisons of continuous variables are performed using t-tests or, in the case of skewed variables, using the non-parametric tests. In the multivariate model, the effects of possible confounding factors are considered.

Project personnel Professor Kirsi Sipilä, Research Unit of Population Health, University of Oulu, and Oulu University Hospital (North Ostrobothnia Wellbeing Services County) DDS, PhD Abhishekhi Shrestha, Post Doctoral Researcher, Oulu University Hospital (North Ostrobothnia Wellbeing Services County) (grant researcher) DDS, PhD Marco Antonios Dias da Silva, Post Doctoral Researcher, Research Unit of Population Health, University of Oulu Docent Ritva Näpänkangas, Research Unit of Population Health, University of Oulu, and Oulu University Hospital (North Ostrobothnia Wellbeing Services County) Prof. Mikko Tulppo, Research Unit of Biomedicine and Internal Medicine, University of Oulu PhD, Post Doctoral researcher Rasmus Valtonen, Research Unit of Biomedicine and Internal Medicine, University of Oulu DDS, PhD Student Elina Heikkinen, Finnish Student Health Service, Oulu, and University of Oulu.

PhD Student Niklas Kakko, University of Oulu PhD Student Riikka Hauru, University of Oulu Prof. Minna Isomursu, Digital Health, University of Oulu DDS, PhD Taina Kankaala, University of Oulu and Well-being Services of North Osthrobotnia County Collaborators DDS, PhD Outi Huhtela, Unit of Dentistry, Faculty of Health Sciences, University of Eastern Finland, and Kuopio University Hospital.

Prof. Em. Martti T. Tuomisto, Clinical psychology and psychotherapist training, Faculty of Social Sciences (Psychology), University of Tampere MD, PhD Juha Markkula, Sleep and Breathing Center, Turku University Hospital and University of Turku, Department of Psychiatry Psychologist Vuokko Hägg, Private practice, Espoo. DDS, PhD, senior dentist Viivi Alaraudanjoki, Finnish Student Health Service, Oulu

Responsible science For the pilot study and clinical trial, ethical permission has been obtained from the Ethics Committee of the North Ostrobothnia Wellbeing Services county (#1/2024). Participation in the study is voluntary, and the subjects are asked to provide a written consent. Subjects have the right to refuse participation at all phases of the study. The subjects are informed about the findings of the study. Data is disclosed to investigators without personal identification number, meaning that individual investigators are not aware of the subject's identity. Due to the General Data Protection Regulation (GDPR), the data is saved in a protected file on the server of University of Oulu. Furthermore, University of Oulu has currently intellectual property rights for Relappy.

The research promotes open science; results are presented in national and international congresses. More publicity will also be gained through publications in media. The results will be published in high impact, open access journals of dentistry or medicine. According to the University publishing policy, all reports are available for public access. Published articles will be stored to the University of Oulu open access repository Jultika. The possible theses from the project will be published in the University of Oulu series.

The project will generate more well-being and contribute to the quality of life for the people. It also promotes equality in health by offering the AR program for wider use. Development of cost-effective prevention and intervention might create equal prospects in terms of health and functional capacity.

In recruitment, equality issues are given special attention. In the research group, gender equality is well realised. The project will promote sustainability. Use of Relappy is expected to decrease the use of materials and medications that are used for pain conditions. For example, occlusal splint, which is a usual treatment method for TMD, is made of plastic material. If Relappy replaces the splint treatment at least partly, it will reduce plastic waste as well as the use of other materials, such as silicon and alginate, that are used as impression material in the fabrication process. The use of Relappy also eliminates paper material as the instructions and exercise diary are saved in electronic format.

ELIGIBILITY:
Inclusion Criteria:

* presence of TMD pain diagnosis (myalgia, myofascial pain with referral, arthralgia and/or headache attributed to TMD), based on validated, international Diagnostic Criteria for TMD Axis I criteria
* the patient has a full dentition (lack of a single tooth in a balanced occlusion does not preclude participation)

Exclusion Criteria:

* serious general illnesses such as rheumatism, schizophrenia or other serious mental illness
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
TMD pain-related intensity | from baseline until 1 year from baseline
  The patient fill in a webropol-based questionnaire on Graded Chronic Pain Scale (GCPS2.0) included in the validated Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). The data is collected at baseline and at the 6-week, 3-month and 1-year follow-up points (after beginning the treatment). Mean pain-related intensity is mean of current, worst and average intensity of pain (on a scale from 0 (no pain) to 10 (worst pain).
TMD pain-related interference | from baseline until 1 year from baseline
  The patient fill in a webropol-based questionnaire on Graded Chronic Pain Scale (GCPS2.0) included in the validated Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). The data is collected at baseline and at the 6-week, 3-month and 1-year follow-up points (after beginning the treatment). The mean pain-related interference (during preceding 30 days) is calculated as mean of interference on daily activities, social activities and ability to work, using a scale from 0 (no interference) to 10 (unable to carry on any activities).

SECONDARY OUTCOMES:
Body pain symptoms | From baseline until 1 year after baseline
  The patient fill in a webropol-based questionnaire on body pain symptoms. Number of body pain sites is calculated (from 0 to 9 pain sites). The data is collected at baseline and at the 6-week, 3-month and 1-year follow-up points (after beginning the treatment).
Depression symptoms | from baseline until 1 year after baseline
  Questions on depression symptoms are included in the webropol-based questionnaire. They are assessed with the validated DC/TMD Axis II questionnaire Patient Health Questionnaire-9 (PHQ-9). A sum score is calculated, using a scale from 0 (no symptoms) to 27 (highest number of symptoms). The data is collected at baseline and at the 6-week, 3-month and 1-year follow-up points (after beginning the treatment).
Physical symptoms | from baseline until 1 year after baseline
  Questions on unspecific physical symptoms are included in the webropol-based questionnaire. They are assessed with the validated DC/TMD Axis II Patient Health Questionnaire-15 (PHQ-15). A sum score is calculated, using a scale from 0 (no symptoms) to 30 (highest number of symptoms). The data is collected at baseline and at the 6-week, 3-month and 1-year follow-up points (after beginning the treatment).
Anxiety symptoms | from baseline until 1 year after baseline
  Questions on anxiety symptoms are included in the webropol-based questionnaire. They are assessed with the validated DC/TMD Axis II anxiety symptoms questionnaire (General Anxiety Disorder-7, GAD-7). The total sum score ranges from 0 (no anxiety) to 21 (the most severe symptoms). The data is collected at baseline and at the 6-week, 3-month and 1-year follow-up points (after beginning the treatment).
Sleep quality | from baseline until 1 year after baseline
  Sleep quality is measured with a validated SCI (Sleep Condition Indicator) questionnaire (in webropol, at baseline and 6 weeks, 3 months and 1 year after baseline). A total score (ranging from 0 to 32) is calculated, with higher scores indicating better sleep. A score of 16 or less may suggest insomnia.
Sleep diary | from baseline until 1 year after baseline
  Sleep diary is registered in Oneiros application (Oneiros Therapies Ltd). The diary includes data (for every night) on sleeping time (minutes), latency in falling asleep (minutes), number of arousal times, total duration of arousals (minutes) and self-estimated quality of sleep (on a scale 0 to 10, the higher number indicating better quality). The data is collected for 2 weeks before treatment and at 3-month and 1-year follow-ups.
Heart rate variability | from baseline until 1 year after baseline
  A sub-sample (n=62) is formed from the patients from Oulu for whom measurements of ANS activity are made before the treatment and 3 months and 1 year after beginning of the treatment. Heart rate variability (HRV) is measured. HRV is a continuous variable. Lower value refers to weaker autonomic nervous system system function.
Baroreflex sensitivity (BRS) | from baseline until 1 year after baseline
  A sub-sample (n=62) is formed from the patients from Oulu for whom measurements of ANS activity are made before the treatment and 3 months and 1 year after beginning of the treatment. Baroreflex sensitivity (BRS) is measured. BRS is a continuous variable. Lower values refer to weaker autonomic nervous system system function.
Body composition (Inbody) | from baseline until 1 year after baseline
  A sub-sample (n=62) is formed from the patients from Oulu for whom measurements of ANS activity are made before the treatment and 3 months and 1 year after beginning of the treatment. Body composition is measured (InBody 720, InBody Co. Korea). The index describes the weight (kg)/muscle mass/fat mass. Value from 70 to 90 means normal, and value 90 or more means muscular.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Undecided
All data contains sensitive information and is protected by local and EU legislation about data security and scientific research (EU General Data Protection Regulation 2016/679, articles 6, 1e and 9, 2i). The data is available on reasonable request from the PI and with permission of University of Oulu.

REFERENCES:
- [Background] Hietaharju M, Napankangas R, Sipila K, Teerijoki-Oksa T, Tanner J, Kemppainen P, Tolvanen M, Suvinen T. Importance of the Graded Chronic Pain Scale as a Biopsychosocial Screening Instrument in TMD Pain Patient Subtyping. J Oral Facial Pain Headache. 2021 Fall;35(4):303-316. doi: 10.11607/ofph.2983. PMID 34990499
- [Background] Huhtela OS, Napankangas R, Suominen AL, Karppinen J, Kunttu K, Sipila K. Association of psychological distress and widespread pain with sympatoms of temporomandibular disorders and self-reported bruxism in students. Clin Exp Dent Res. 2021 Dec;7(6):1154-1166. doi: 10.1002/cre2.472. Epub 2021 Jul 20. PMID 34289266
- [Background] Hayes-Skelton SA, Usmani A, Lee JK, Roemer L, Orsillo SM. A Fresh Look at Potential Mechanisms of Change in Applied Relaxation for Generalized Anxiety Disorder: A Case Series. Cogn Behav Pract. 2012 Aug;19(3):451-462. doi: 10.1016/j.cbpra.2011.12.005. PMID 23888107
- [Background] Kemani MK, Hesser H, Olsson GL, Lekander M, Wicksell RK. Processes of change in Acceptance and Commitment Therapy and Applied Relaxation for long-standing pain. Eur J Pain. 2016 Apr;20(4):521-31. doi: 10.1002/ejp.754. Epub 2015 Dec 18. PMID 26684472
- [Background] Espie CA, Kyle SD, Hames P, Gardani M, Fleming L, Cape J. The Sleep Condition Indicator: a clinical screening tool to evaluate insomnia disorder. BMJ Open. 2014 Mar 18;4(3):e004183. doi: 10.1136/bmjopen-2013-004183. PMID 24643168
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Huhtela OS, Koivisto N, Hagg V, Sipila K. Effectiveness of applied relaxation method vs splint in treatment of temporomandibular disorders in Finnish students. J Oral Rehabil. 2020 Feb;47(2):123-131. doi: 10.1111/joor.12884. Epub 2019 Nov 9. PMID 31493297
- See also: Researcher profile of Kirsi Sipilä/ University of Oulu, Finland — https://www.oulu.fi/en/researchers/kirsi-sipila